CLINICAL TRIAL: NCT03459963
Title: Risks and Benefits of Urinary Catheterization in Elective Cesarean Section: A Randomized Controlled Trial
Brief Title: Risks and Benefits of Urinary Catheter in Elective Cesarean Section
Acronym: catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Dina Islam, Doctor, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: elgammal
Record Dates: First submitted 2018-02-28; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Urinary Catheterization
Keywords: catheter; cesarean section; urinary tract infection; patient's satisfaction
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group C (Experimental): indwelling urinary catheter
  Interventions: Device: indwelling urinary catheter
- group N (No Intervention): Non cathetrized patients

INTERVENTIONS:
Device: indwelling urinary catheter — 85 women undergoing first elective CS will be catheterized immediately preoperatively using Foley's catheter by applying catheterization precautions.
  Arms: group C

SUMMARY:
This study aims to compare the routine use versus non-use of urethral catheterization in women undergoing first elective cesarean section as regard to intraoperative and postoperative complications

DETAILED DESCRIPTION:
This randomized controlled trial will be done at Ain Shams University Maternity One hundred and seventy pregnant women scheduled for first elective CS attending at outpatient clinic will be chosen after complete history and physical examination to determine eligibility for inclusion after taking their consent with full explanation of the study including potential benefits and risks.

The study population will be randomized using computer sequence program in 1:1 ratio. Allocation of every patient to one of the studied groups will be done using opaque envelops.

The studied groups will be either Group C or Group N For both groups

* A written consent will be taken.
* Full history to exclude medical problems that need special care.
* Full history to exclude UTI or recurrent UTI during pregnancy.
* A single dose of 2 gm cefazolin will be given IV pre-incision for preoperative antibiotic prophylaxis (Sullivan et al., 2007).
* midstream urine samples will be collected preoperative to exclude UTI and 24 hours postoperatively after giving the instructions to the patients (washing hands and genitals ,pass some urine into the toilet then without stopping catch some urine in a sterile container ) to be analyzed for presence of UTI

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing first elective CS at term pregnancy (37-41w gestation).
* haemodynamically stable

Exclusion Criteria:

* History of recurrent UTI during pregnancy, current UTI
* presence of Medical complications that requiring special care e.g: diabetes with pregnancy, hypertensive disorders with pregnancy, cardiac disease, chronic renal disease,
* previous cesarean section
* Previous abdominal surgery which may be associated with extensive adhesions, -polyhydraminos
* fetal macrosomia
* significant vaginal bleeding
* Contraindication for the antibiotic used e.g: anaphylaxis
* Need for extensive use of antibiotics more than the prophylactic dose
* Spinal anesthesia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 170 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Presence of UTI | 24-h postoperative
  midstream urine samples were collected 24 hours postoperatively after giving the instructions to the patients and tested for presence of UTI. These fresh non-centrifuged urine samples were collected and tested for leukocyte esterase and nitrite using (Convergys urine matrix 10, Germany) strips. Nitrite will be considered positive if there is change in color of dipstick from colorless towards pink within 60 seconds. Leukocyte esterase will be considered positive if there is change in color from off-white towards purple within 2 minutes

SECONDARY OUTCOMES:
Operative duration | intraoperative
  The time taken for surgery from skin opening to complete skin closure,
Bladder injury incidence. | intraoperative
  accidental bladder injury during operation
Intraoperative need of urethral catheter in N group | intraoperative
  intraoperative need of catheter for any reason
Ambulation time | intraoperative
  from intraoperative skin opening time till the patient is able to move.
Postpartum hemorrhage | first postoperative day
  identified when there is costant trickling f blood or repeated soakage of valval pad within 5 minutes
Urinary retention | first postoperative day
  defined as no spontaneous micturition >24 hours after cesarean delivery
Patient satisfaction | second postoperative day morning
  using four point likert scale from 1-4 (as 1 = not satisfied, 2 = partial satisfied, 3 = satisfied, 4 = very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Tamer F borg, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital., Cairo, Egypt